CLINICAL TRIAL: NCT01363869
Title: Effects of Green Tea on Level of Serum Uric Acid in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kanon Jatuworapruk, Kanon Jatuworapruk M.D, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-11-02-07-13-X
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Hyperuricemia; Gout
Keywords: hyperuricemia; gout; uric acid; xanthine oxidase inhibitor; green tea; catechins; antioxidant
MeSH Terms: conditions — Hyperuricemia; Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Green tea extracts 2 gm/day (Experimental): Green tea extracts 2 gm/day for 14 days
  Interventions: Dietary Supplement: green tea extracts 2 gm/day
- Green tea extracts 4 gm/day (Experimental): Green tea extracts 4 gm/day for 14 days
  Interventions: Dietary Supplement: green tea extracts 4 gm/day
- Green tea extracts 6 gm/day (Experimental): Green tea extracts 6 gm/day for 14 days
  Interventions: Dietary Supplement: green tea extracts 6 gm/day

INTERVENTIONS:
Dietary Supplement: green tea extracts 2 gm/day — Green tea extracts capsule (1 gm per capsule), taken after meal, twice daily for 14 days.
  Total dosage is 2 grams per day.
  Arms: Green tea extracts 2 gm/day
Dietary Supplement: green tea extracts 4 gm/day — Green tea extracts capsule (1 gm per capsule), taken after meal, twice daily for 14 days.
  Total dosage is 4 grams per day.
  Arms: Green tea extracts 4 gm/day
Dietary Supplement: green tea extracts 6 gm/day — Green tea extracts capsule (1 gm per capsule), taken after meal, twice daily for 14 days.
  Total dosage is 6 grams per day.
  Arms: Green tea extracts 6 gm/day

SUMMARY:
Green tea has been extensively investigated for several potential health benefits. Previous studies have suggested that green tea may lower serum uric acid level in human. The purpose of this study is to investigate uric-lowering properties of green tea in healthy individuals.

DETAILED DESCRIPTION:
Elevated serum uric acid is related to the risk of development of gout, the most common inflammatory arthritis in men. Allopurinol, a xanthine oxidase inhibitor, is one of the uric-lowering agents commonly used in patients suffering from recurrent and chronic gout. Nevertheless, its use is limited by adverse effects and serious allergic reaction in some patients.

Green tea is one of the most frequently consumed beverages, particularly in Japan. Green tea contains high level of catechins, in which Epigallocatechin gallate (EGCG) is the most abundant compound among other types of catechins. Antioxidant effect contributes to various potential health benefits of green tea. Several in-vitro studies have found that green tea inhibits xanthine oxidase activity and subsequently decreases reactive oxygen species (ROS) and uric acid production. We therefore would like to investigate the hypouricemic effects of green tea.

The study consists of three periods with a total duration of four weeks. The first week is the control period. The following two weeks is the interventional period and the last week is the follow up period. Thirty healthy participants will be randomly assigned into three experimental groups, receiving 2 gm/day, 4 gm/day and 6 gm/day (in capsule, two times after meal) of green tea extract during interventional period. Blood and urine samples will be taken at the beginning and at the end of each study period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Healthy individuals
* Normal renal and liver function from blood tests

Exclusion Criteria:

* Presence of co-morbidity or currently ill
* Currently using any medication or nutritional supplement product that may affect serum uric acid level
* Serum creatinine higher than 1.5 mg/dl
* Abnormal serum Aspartate aminotransferase (AST) and/or Alanine transaminase (ALT)
* Greater than 15% change in serum uric acid during control period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
serum uric acid | 4 weeks (prior to, immediately after and 7 days after intervention)

SECONDARY OUTCOMES:
urinary uric acid excretion | 4 weeks (prior to, immediately after and 7 days after intervention)
serum antioxidant activity | 4 weeks (prior to, immediately after and 7 days after intervention)
serum EGCG level | 1 week (immediately after and 7 days after intervention)
  Measurements of serum level of epigallocatechin gallate (EGCG)
Adverse events | 4 week (prior to, immediately after and 7 days after intervention)
  Adverse events during 4-week study

CONTACTS AND LOCATIONS:
Overall Officials: Kanon Jatuworapruk, M.D, Principal Investigator — Department of Internal medicine, Faculty of Medicine, Chiang Mai University, Thailand
Locations (1):
- Department of Internal Medicine, Faculty of Medicine, Chiang Mai University, Chiang Mai, Chiang Mai, Thailand